CLINICAL TRIAL: NCT00053898
Title: A Clinical Trial Comparing Anastrozole With Tamoxifen in Postmenopausal Patients With Ductal Carcinoma in Situ (DCIS) Undergoing Lumpectomy With Radiation Therapy
Brief Title: Anastrozole or Tamoxifen in Treating Postmenopausal Women With Ductal Carcinoma in Situ Who Are Undergoing Lumpectomy and Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network); American College of Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSABP B-35; NSABP-B-35; SWOG-NSABP-B-35; NCCTG-NSABP-B-35; ACOSOG-NSABP-B-35
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Anastrozole; Tamoxifen; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): tamoxifen 20 mg/day and an anastrozole look-alike placebo for 5 years
  Interventions: Drug: tamoxifen citrate; Radiation: Radiation Therapy
- Group 2 (Experimental): anastrozole, 1 mg/day and an tamoxifen look-alike placebo for 5 years
  Interventions: Drug: anastrozole; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: anastrozole — 1 mg/day and placebo for 5 years
  Arms: Group 2
Drug: tamoxifen citrate — 20 mg/day and placebo for 5 years
  Arms: Group 1
Radiation: Radiation Therapy — Adjuvant radiation therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Tamoxifen may fight breast cancer by blocking the use of estrogen. Anastrozole may fight breast cancer by decreasing estrogen production. It is not yet known whether anastrozole is more effective than tamoxifen in preventing the recurrence of breast cancer.

PURPOSE: This randomized phase III trial is studying anastrozole to see how well it works compared to tamoxifen in preventing the recurrence of breast cancer in postmenopausal women with ductal carcinoma in situ who are undergoing lumpectomy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the value of anastrozole vs tamoxifen, in terms of preventing recurrence (i.e., local, regional, and distant recurrences and contralateral breast cancer), after lumpectomy and radiotherapy in postmenopausal women with ductal carcinoma in situ (DCIS).
* Compare subsequent disease occurrence, in terms of invasive breast cancer (local, regional, distant, or contralateral), ipsilateral and contralateral breast cancer (invasive and DCIS), and non-breast second primary malignancies, in patients treated with these drugs.
* Compare quality of life and symptoms of patients treated with these drugs.*
* Compare quality-adjusted survival time of patients treated with these drugs.*
* Compare the occurrence of osteoporotic fractures in patients treated with these drugs.
* Compare disease-free and overall survival of patients treated with these drugs. NOTE: *The quality of life study closed to accrual as of 12/28/04.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (under 60 vs 60 and over). Patients are randomized to 1 of 2 treatment arms (arm I and arm II closed to accrual as of 6/15/06).

* Arm I (closed to accrual as of 6/15/06): Patients receive oral tamoxifen and oral placebo once daily for 5 years.
* Arm II (closed to accrual as of 6/15/06): Patients receive oral anastrozole and oral placebo once daily for 5 years.

Beginning within 8 weeks of randomization, all patients also undergo whole breast radiotherapy, unless the patient is enrolled in protocol NSABP-B-39 and randomized to the partial breast irradiation group.

Patients are followed every 6 months for 5 years, and then annually thereafter.

For patients enrolled in the quality of life study, quality of life is assessed at baseline and then every 6 months for 6 years.*

NOTE: *The quality of life study closed to accrual as of 12/28/04.

PROJECTED ACCRUAL: A total of 3,000 patients (1,500 per treatment arm) will be accrued for this study within 5 years (arm I and arm II closed to accrual as of 6/15/06).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS) of the breast

  * Mixed DCIS and lobular carcinoma in situ (LCIS) allowed
* Must have undergone lumpectomy

  * Margins must be histologically free of disease
  * Re-excision to obtain tumor-free margins allowed
  * No more than 84 days since prior lumpectomy or re-excision
* More than 1 area of DCIS allowed provided all disease is removed with tumor-free margins

  * Masses or clusters of calcification that are clinically or mammographically suspicious must be biopsied
* No prior invasive breast cancer or DCIS

  * Patients with a history of LCIS are eligible
* No prior or concurrent invasive (including microinvasive) breast cancer

  * DCIS "suspicious" for microinvasion allowed
* No bilateral malignancy

  * No mass or mammographic abnormality suspicious for malignancy in the opposite breast unless not malignant as proven by biopsy
* No Paget's disease of the nipple
* No positive ipsilateral axillary or intramammary nodes

  * No palpable nodes in the ipsilateral or contralateral axilla or palpable supraclavicular or infraclavicular nodes unless not involved with tumor as proven by biopsy
* Hormone receptor status:

  * Estrogen- or progesterone-receptor positive as determined by immunohistochemistry

    * Borderline results are considered positive

PATIENT CHARACTERISTICS:

Age

* See Menopausal status

Sex:

* Female

Menopausal status:

* Postmenopausal as defined by at least 1 of the following:

  * Prior documented bilateral oophorectomy
  * At least 12 months without spontaneous bleeding
  * Age 55 or over with prior hysterectomy without oophorectomy
  * Age 54 or under with prior hysterectomy without oophorectomy with a documented follicle-stimulating hormone level in the postmenopausal range

Performance status

* Zubrod 0-2

Life expectancy

* At least 10 years (excluding diagnosis of breast cancer)

Hematopoietic

* WBC normal

Hepatic

* AST normal
* Bilirubin normal
* Alkaline phosphatase normal
* No hepatic disease that would preclude administration of study drugs

Renal

* Creatinine normal
* No renal disease that would preclude administration of study drugs

Cardiovascular

* No prior documented cerebral vascular accident or transient ischemic attack
* No prior deep vein thrombosis
* No cardiovascular disease that would preclude administration of study drugs
* No uncontrolled hypertension (i.e., systolic blood pressure at least 180 mm Hg or diastolic blood pressure at least 110 mm Hg based on the average of 2 or more readings at each of 2 or more visits after initial screening)
* No uncontrolled atrial fibrillation

Pulmonary

* No pulmonary embolus

Other

* Not pregnant or nursing
* Patients with a history of non-breast malignancies are eligible provided they have been disease-free for ≥ 5 years and are deemed by their physician to be at low risk for recurrence
* No other malignancy within the past 5 years except treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, carcinoma in situ of the colon, or melanoma in situ
* No psychiatric or addictive disorders that would preclude informed consent
* No uncontrolled diabetes, defined as hemoglobin A1C greater than 9% (fasting glucose 200 mg/dL)
* No nonmalignant systemic disease that would preclude administration of study drugs

PRIOR CONCURRENT THERAPY:

Endocrine therapy

* No prior or concurrent aromatase inhibitors (e.g., exemestane or letrozole) or tamoxifen
* No concurrent raloxifene or other selective estrogen receptor modulators
* No concurrent sex hormone therapy (e.g., estrogen or progesterone replacement therapy, oral contraceptives, androgens, luteinizing hormone releasing hormone analogs, prolactin inhibitors, or antiandrogens)

  * Low-dose estrogen vaginal creams or Estring allowed

Radiotherapy

* Radiotherapy for this cancer initiated before study is allowed

Surgery

* See Disease Characteristics
* No prior or concurrent mastectomy for DCIS
* Prior sentinel node biopsy or axillary node dissection allowed provided nodes are pathologically negative

Other

* No concurrent warfarin
* No other systemic therapy for this cancer initiated before study
* No other concurrent anticancer therapy unless permitted by the protocol investigator
* No concurrent participation in another clinical trial of therapy for DCIS

  * Concurrent participation in protocol NSABP-B-39 allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3104 (Actual)
Dates: Start 2003-01; Primary Completion 2015-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (740):
- United States (724):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - East Alabama Medical Center, Opelika, Alabama
  - Cancer Center at Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Saint Joseph's Mercy Cancer Center, Hot Springs, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Washington Township Hospital, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Saint Rose Hospital, Hayward, California
  - Stevens Cancer Center at Scripps Memorial Hospital, La Jolla, California
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Pacific Shores Medical Group Comprehensive Hematology-Oncology Services - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Memorial Medical Center Cancer Services, Modesto, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Care Medical Center, Pleasanton, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Torrance Memorial Medical Center, Torrance, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Ruby L. Golleher Cancer Program at Presbyterian Intercommunity Hospital, Whittier, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Watson Clinic, LLC, Lakeland, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Robert and Carol Weissman Cancer Center at Martin Memorial, Stuart, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Portneuf Cancer Center at Portneuf Medical Center, Pocatello, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Medical and Surgical Specialists, L L C, Galesburg, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Wasser Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Regional Cancer Institute at Bloomington Hospital, Bloomington, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Methodist Cancer Center at Clarian Health, Indianapolis, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Community Hospital, Munster, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, P.C. - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Lexington Clinic Cancer Center, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisville Oncology at Norton Cancer Center, Louisville, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Cancer Treatment Center at Christus Schumpert St. Mary Place, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - MaineGeneral Medical Center - Waterville Campus, Waterville, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - St. Mary's Hospital, Leonardtown, Maryland
  - Kaiser Permanente Capital Area Medical Group - Shady Grove Facility, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital, Fall River, Massachusetts
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Franklin Medical Center, Greenfield, Massachusetts
  - Lawrence Memorial Hospital of Medford, Medford, Massachusetts
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Commonwealth Hematology-Oncology P. C. - Quincy, Quincy, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Hospital, Pontiac, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Carson-Tahoe Cancer Services at Carson Tahoe Regional Healthcare, Carson City, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Parkland Oncology-Hematology Clinic at Parkland Medical Center, Derry, New Hampshire
  - Seacoast Cancer Center at Wentworth-Douglass Hospital, Dover, New Hampshire
  - Exeter Hospital Center for Cancer Care, Exeter, New Hampshire
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Capital Health System Regional Cancer Center, Trenton, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - South Jersey Healthcare Regional Cancer Center, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Underwood Memorial Hospital, Woodbury, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Lovelace Medical Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Santa Fe Cancer Center at St. Vincent Hospital, Santa Fe, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Amsterdam Community Cancer Program, Amsterdam, New York
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology, P.C. at Cavell Cancer Treatment Program, Hudson, New York
  - New York Oncology Hematology, P.C., Latham, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Union State Bank Cancer Center at Nyack Hospital, Nyack, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Riverview Cancer Care Medical Associates, PC, Rexford, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Genesee Surgical Associates - Linden Oaks Medical Campus, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - New York Oncology Hematology, P.C. - Ellis Office, Schenectady, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - St. Joseph's Hospital Health Center - Syracuse, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Samaritan Hospital at Northeast Health, Troy, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Cancer Treatment Center at Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care, Incorporated - Blue Ash, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Huron Hospital Cancer Care Center, Cleveland, Ohio
  - Euclid Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - St. Joseph Cancer Center at St. Joseph Health Center, Warren, Ohio
  - South Pointe Hospital Cancer Care Center, Warrensville Heights, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Comanche County Memorial Hospital, Lawton, Oklahoma
  - Integris Oncology Services, Oklahoma City, Oklahoma
  - Mercy Health Center, Oklahoma City, Oklahoma
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, P.C. at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Richard G. Laube Cancer Center at Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Meadville Medical Center, Meadville, Pennsylvania
  - Cancer Center at Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Frankford Hospital - Torresdale Campus, Philadelphia, Pennsylvania
  - Chestnut Hill Healthcare Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Wellspan Health, York, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Cancer Care Institute of Carolina at Aiken Regional Medical Centers, Aiken, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Erlanger Cancer Center, Chattanooga, Tennessee
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Centers for Cancer Care, Memphis, Tennessee
  - Seton Shivers Cancer Program at Brackenridge Hospital, Austin, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Mount Ascutney Hospital, Windsor, Vermont
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Rappahannock General Hospital, Kilmarnock, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Overlake Cancer Center at Overtake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Providence Centralia Hospital Regional Cancer Center, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - St. Mary Regional Cancer Center at St. Mary Medical Center, Walla Walla, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Fox Valley Surgical Associates at Appleton Medical Center, Appleton, Wisconsin
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Fish Hatchery, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - St. Joseph Regional Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at All Saints Medical Center, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconsin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (13):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Ambulatory Care Center at Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - CHUM Hopital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- Puerto Rico (3):
  - Andres Grillasca Hospital, Ponce
  - Hato Rey Hematology/Oncology Group, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Background] Land SR, Ritter MW, Costantino JP, Julian TB, Cronin WM, Haile SR, Wolmark N, Ganz PA. Compliance with patient-reported outcomes in multicenter clinical trials: methodologic and practical approaches. J Clin Oncol. 2007 Nov 10;25(32):5113-20. doi: 10.1200/JCO.2007.12.1749. PMID 17991930
- [Background] Margolese RG, Cecchini RS, Julian TB, Ganz PA, Costantino JP, Vallow LA, Albain KS, Whitworth PW, Cianfrocca ME, Brufsky AM, Gross HM, Soori GS, Hopkins JO, Fehrenbacher L, Sturtz K, Wozniak TF, Seay TE, Mamounas EP, Wolmark N. Anastrozole versus tamoxifen in postmenopausal women with ductal carcinoma in situ undergoing lumpectomy plus radiotherapy (NSABP B-35): a randomised, double-blind, phase 3 clinical trial. Lancet. 2016 Feb 27;387(10021):849-56. doi: 10.1016/S0140-6736(15)01168-X. Epub 2015 Dec 11. PMID 26686957
- [Background] Ganz PA, Cecchini RS, Julian TB, Margolese RG, Costantino JP, Vallow LA, Albain KS, Whitworth PW, Cianfrocca ME, Brufsky AM, Gross HM, Soori GS, Hopkins JO, Fehrenbacher L, Sturtz K, Wozniak TF, Seay TE, Mamounas EP, Wolmark N. Patient-reported outcomes with anastrozole versus tamoxifen for postmenopausal patients with ductal carcinoma in situ treated with lumpectomy plus radiotherapy (NSABP B-35): a randomised, double-blind, phase 3 clinical trial. Lancet. 2016 Feb 27;387(10021):857-65. doi: 10.1016/S0140-6736(15)01169-1. Epub 2015 Dec 11. PMID 26686960
- [Derived] Duggal S, Robin J, Julian TB. Ductal carcinoma in situ: an overview. Expert Rev Anticancer Ther. 2013 Aug;13(8):955-62. doi: 10.1586/14737140.2013.820557. PMID 23984897

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Tamoxifen + Anastrozole Placebo: tamoxifen 20 mg/day and an anastrozole look-alike placebo for 5 years
  tamoxifen citrate: 20 mg/day and placebo for 5 years
  Radiation Therapy: Adjuvant radiation therapy
- Group 2: Anastrozole + Tamoxifen Placebo: anastrozole, 1 mg/day and an tamoxifen look-alike placebo for 5 years
  anastrozole: 1 mg/day and placebo for 5 years
  Radiation Therapy: Adjuvant radiation therapy
Period: Overall Study
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Started | 1552 | 1552
Completed | 1538 | 1539
Not Completed | 14 | 13
Not completed — No follow-up data from any source | 9 | 12
Not completed — Follow-up from telephone contact only | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Tamoxifen + Anastrozole Placebo: tamoxifen 20 mg/day and an anastrozole look-alike placebo for 5 years
  Drug: tamoxifen citrate
  20 mg/day and placebo for 5 years
  Radiation: Radiation Therapy
  Adjuvant radiation therapy
- Group 2: Anastrozole + Tamoxifen Placebo: anastrozole, 1 mg/day and an tamoxifen look-alike placebo for 5 years
  Drug: anastrozole
  1 mg/day and placebo for 5 years
  Radiation: Radiation Therapy
  Adjuvant radiation therapy
- Total: Total of all reporting groups
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo | Total
Number analyzed (Participants) | 1552 | 1552 | 3104
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (7.8) | 61.1 (7.8) | 61.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1552 | 1552 | 3104
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Free From Breast Cancer
Description: Percentage of patients free from breast cancer event at 10 years where events include local, regional, or distant recurrence or contralateral breast cancer, invasive or DCIS.
Time Frame: 10 years
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
percentage of participants event-free | 89.1 | 93.1

2. Secondary Outcome: Percentage of Patients Free From Invasive Breast Cancer
Description: Percentage of patients free from an invasive breast cancer event where events include invasive local, regional, or distant recurrence, or contralateral breast cancer, occurring as a first cancer event. Note that this endpoint includes only invasive breast cancers and the primary endpoint includes both invasive and DCIS breast cancers.
Time Frame: 10 years
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
percentage of participants event-free | 93.3 | 96.4

3. Secondary Outcome: Percentage of Patients Free From Ipsilateral Recurrence
Description: Percentage of patients free from a breast cancer recurrence in the ipsilateral breast (invasive and DCIS), occurring as a first cancer event.
Time Frame: 10 years
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
percentage of participants event-free | 94.6 | 96.4

4. Secondary Outcome: Percentage of Patients Free From Contralateral Breast Cancer
Description: Percentage of patients free from a breast cancer recurrence in the contralateral breast (invasive and DCIS), occurring as a first cancer event.
Time Frame: 10 years
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
percentage of participants event-free | 94.7 | 97.0

5. Secondary Outcome: Percentage of Patients Free From Non-breast Secondary Cancer
Description: Percentage of patients free from any non-breast second primary cancer other than squamous or basal cell carcinoma of the skin, carcinoma in situ of the colon, melanoma in situ, or carcinoma in situ of the cervix, occurring as a first cancer event.
Time Frame: 10 years
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
percentage of participants event-free | 91.5 | 91.9

6. Secondary Outcome: Percentage of Patients Free From Osteoporotic Fractures
Description: Percentage of patients free from fractures of the hip, spine, and wrist.
Time Frame: 10 years
Population: The analysis for osteoporotic fractures included those whose method of contact for follow-up was by telephone. Two participants were excluded from the analysis because their date of fracture was unknown.
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1542 | 1539
percentage of participants event-free | 96.0 | 95.3

7. Secondary Outcome: Percentage of Patients Alive and Disease-free
Description: Percentage of patients free from a disease-free survival event where events include any recurrence, second primary cancer, and death from any cause. Lobular carcinoma in situ (LCIS), basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the colon, melanoma in situ, and cervical carcinoma in situ will not be included as recurrences or second primary cancer.
Time Frame: 10 years
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
percentage of participants event-free | 77.9 | 82.7

8. Secondary Outcome: Percentage of Patients Alive (Overall Survival)
Description: Percentage of patients alive.
Time Frame: 10 years
Population: The analysis for overall survival included those whose method of contact for follow-up was by telephone.
Measure: Number; unit: percentage of participants event-free
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1543 | 1540
percentage of participants event-free | 92.1 | 92.5

9. Secondary Outcome: Quality of Life-Short Form 12 (SF-12) Physical Health Component Score
Description: The primary outcome of the QOL substudy was the Medical Outcomes Study-Short Form 12 (SF-12) physical health component scale score. The SF-12 physical score was calculated to have a range of 0-100 and was normalized to have a mean of 50 and a standard deviation of 10 in the general population. Higher scores indicate better health.
Time Frame: 5 years
Population: The Quality of Life study was performed in a subset of B-35 participants. Participants were required to have submitted a baseline and at least one follow-up QOL form to be included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 601 | 592
units on a scale | 46.20 (10.13) | 45.38 (10.25)

10. Secondary Outcome: Quality-adjusted Survival Time
Description: The mean quality-adjusted survival time (in months) in each treatment group, estimated by the Quality-Adjusted Time without Symptoms and Toxicity (Q-TWIST) method.
Time Frame: 10 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrozole + Tamoxifen Placebo
Number analyzed (Participants) | 1538 | 1539
months | 104.4 [101.8 to 106.9] | 102.9 [100.9 to 104.9]

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Groups:
- Group 2: Anastrazole + Tamoxifen Placebo: anastrozole, 1 mg/day and a tamoxifen look-alike placebo for 5 years
  Drug: anastrozole
  1 mg/day and placebo for 5 years
  Radiation: Radiation Therapy
  Adjuvant radiation therapy
Arm/Group | Group 1: Tamoxifen + Anastrozole Placebo | Group 2: Anastrazole + Tamoxifen Placebo
Serious Adverse Events (participants affected / at risk) | 73/1535 | 62/1535
Other Adverse Events (participants affected / at risk) | 1024/1535 | 1064/1535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Tamoxifen + Anastrozole Placebo (N=1535) | Group 2: Anastrazole + Tamoxifen Placebo (N=1535)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 1 | 0
Blood antidiuretic hormone abnormal (Investigations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 3 | 3
Cardiac troponin I increased (Investigations) | 4 | 5
Cardiac troponin T increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 2 | 0
Colitis (Gastrointestinal disorders) | 2 | 1
Confusion (Psychiatric disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
CPK increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 2 | 7
Death NOS (General disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Depression (Psychiatric disorders) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Infections and infestations - Other, specify (Infections and infestations) | 2 | 8
Intracranial hemorrhage (Nervous system disorders) | 3 | 2
Investigations - Other, specify (Investigations) | 1 | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 6 | 8
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 7 | 7
Neuralgia (Nervous system disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0
Platelet count decreased (Investigations) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Stroke (Nervous system disorders) | 1 | 0
Sudden death NOS (General disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 5 | 1
Syncope (Nervous system disorders) | 1 | 2
Thromboembolic event (Vascular disorders) | 20 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 2 | 1
Wound infection (Infections and infestations) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 4 | 0
GGT increased (Investigations) | 0 | 1
Lung infection (Infections and infestations) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 3 | 2
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Tamoxifen + Anastrozole Placebo (N=1535) | Group 2: Anastrazole + Tamoxifen Placebo (N=1535)
Arthralgia (Musculoskeletal and connective tissue disorders) | 358 | 504
Bone pain (Musculoskeletal and connective tissue disorders) | 96 | 152
Cataract (Eye disorders) | 77 | 43
Depression (Psychiatric disorders) | 112 | 126
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 101 | 95
Fatigue (General disorders) | 187 | 196
Headache (Nervous system disorders) | 73 | 86
Hot flashes (Vascular disorders) | 655 | 570
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 124 | 99
Infections and infestations - Other, specify (Infections and infestations) | 216 | 207
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 55 | 91
Myalgia (Musculoskeletal and connective tissue disorders) | 168 | 218
Pain (General disorders) | 78 | 88
Vaginal dryness (Reproductive system and breast disorders) | 137 | 197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days